CLINICAL TRIAL: NCT01400451
Title: A Phase I Trial of Vemurafenib and Ipilimumab in Subjects With V600 BRAF Mutation-positive Metastatic Melanoma
Brief Title: Ph I Ipilimumab Vemurafenib Combo in Patients With v-Raf Murine Sarcoma Viral Oncogene Homolog B1 (BRAF)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: More than 2 of 6 patients treated experienced dose limiting toxicities.
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-161 ST; 2011-000906-22 (EudraCT Number)
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipilimumab + Vemurafenib (Experimental)
  Interventions: Drug: Ipilimumab (BMS-734016); Drug: Vemurafenib

INTERVENTIONS:
Drug: Ipilimumab (BMS-734016) — Injection, intravenous (i.v.), cohort 1: 3 mg/kg, Escalate to cohort 2: 10 mg/kg, Escalate to cohort 3: at Recommended Phase 2 Dose (RP2D), De-escalate cohort 1A: 3 mg/kg, De-escalate cohort -1B: 10 mg/kg, (every three week) Q3wk, upto 2 yrs
  Other Names: Yervoy®; Ipilimumab; BMS-734016
Drug: Vemurafenib — tablets, oral, cohort 1: 960 mg Twice daily (BID) x 28 days after date, cohort 2: 960 mg BID x 28 days after date, cohort 3: at Recommended Phase 2 Dose (RP2D) x 14 days after date, De-escalate cohort 1A: 720 mg BID x 28 days after date, De-escalate cohort -1B: 720 mg BID x 28 days after date , Up to 2 yrs

SUMMARY:
Treatment of subjects who have metastatic melanoma that expresses an activated mutant form of the BRAF oncogene (V600E) with a combination of the specific BRAF inhibitor, Vemurafenib, and the Cytotoxic T Lymphocyte Antigen 4 (CTLA-4) inhibitor mAb Ipilimumab will be safe and feasible and will show preliminary evidence of anti-tumor efficacy and survival in comparison to historical results following treatment with either agent alone.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Metastatic melanoma with activating V600 BRAF mutation
* Measurable Tumor
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1

Exclusion Criteria:

* Autoimmune disease
* Active Brain Metastasis (must be stable after radiation for at least one month)
* Prior therapy with immune stimulating agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - University Of California Los Angeles, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Inst, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Ackerman A, Klein O, McDermott DF, Wang W, Ibrahim N, Lawrence DP, Gunturi A, Flaherty KT, Hodi FS, Kefford R, Menzies AM, Atkins MB, Long GV, Sullivan RJ. Outcomes of patients with metastatic melanoma treated with immunotherapy prior to or after BRAF inhibitors. Cancer. 2014 Jun 1;120(11):1695-701. doi: 10.1002/cncr.28620. Epub 2014 Feb 27. PMID 24577748
- [Derived] Ludlow SP, Pasikhova Y. Cumulative dermatologic toxicity with ipilimumab and vemurafenib responsive to corticosteroids. Melanoma Res. 2013 Dec;23(6):496-7. doi: 10.1097/CMR.0000000000000018. PMID 24025700
- [Derived] Mandala M, Voit C. Targeting BRAF in melanoma: biological and clinical challenges. Crit Rev Oncol Hematol. 2013 Sep;87(3):239-55. doi: 10.1016/j.critrevonc.2013.01.003. Epub 2013 Feb 15. PMID 23415641
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started Nov 2011; Primary Endpoint April 2013; Completed safety follow-up December 2013. Dose-limiting toxicities observed early in dose escalation (Phase I) part of the study. The combination of drugs was not well tolerated, and a maximum tolerable dose was not attained so the study was closed to enrollment and Phase II part was not started.
Pre-assignment Details: 18 participants enrolled; 12 treated with study drug and 6 participants were not treated because they no longer met study criteria. Two of the 12 only received vemurafenib while the other 10 received the combination of vemurafenib and ipilimumab.
Groups:
- 3 mg/kg Ipilimumab + 960 mg Vemurafenib: Lead In Period: 28 Days of 960 mg vemurafenib orally twice daily (starting Day -27 or -13).
  Combination Treatment (Induction of ipilimumab) Period: 3 milligrams per kilogram body weight (mg/kg) ipilimumab intravenously once every 3 weeks for 4 weeks (Week 1, Week 4, Week 7, Week 10) starting on Day 1 plus 960 mg vemurafenib orally twice daily throughout combination treatment.
- 3 mg/kg Ipilimumab + 720 mg Vemurafenib: Lead In Period: 28 Days of 720 mg vemurafenib orally twice daily (starting Day -27 or -13).
  Combination Treatment (Induction of ipilimumab) Period: 3 milligrams per kilogram body weight (mg/kg) ipilimumab intravenously once every 3 weeks for 4 weeks (Week 1, Week 4, Week 7, Week 10) starting on Day 1 plus 720 mg vemurafenib orally twice daily throughout combination treatment.
- 720 mg Vemurafenib: These participants were receiving 720 mg vemurafenib in the Lead in Period prior to starting ipilimumab but after the dose limiting toxicities (DLTs) were identified ipilimumab was not started. Due to disease stabilization, they continued on 720 mg vemurafenib alone orally twice daily. Note: the dose of vemurafenib could be escalated from 720 mg to 960 mg, at the investigator's discretion.
Period: 28 Day Lead In With Vemurafenib Alone
Arm/Group | 3 mg/kg Ipilimumab + 960 mg Vemurafenib | 3 mg/kg Ipilimumab + 720 mg Vemurafenib | 720 mg Vemurafenib
Started | 6 | 4 | 2
Completed | 6 | 4 | 2
Not Completed | 0 | 0 | 0
Period: Combination Treatment (or Intended)
Arm/Group | 3 mg/kg Ipilimumab + 960 mg Vemurafenib | 3 mg/kg Ipilimumab + 720 mg Vemurafenib | 720 mg Vemurafenib
Started | 6 | 4 | 2 (Did not start Ipilimumab but remained on vemurafenib alone.)
Completed | 0 | 0 | 0
Not Completed | 6 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Drug Toxicity | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Disease Progression | 3 | 1 | 1
Not completed — Dose-limiting toxicity | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- 3 mg/kg Ipilimumab + 960 mg Vemurafenib: Lead In Period: 28 Days of 960 mg vemurafenib orally twice daily (starting Day -27 or -13).
  Combination Treatment (Induction of ipilimumab) Period: 3 milligrams per kilogram body weight (mg/kg) ipilimumab intravenously once every 3 weeks for 4 weeks (Week 1, Week 4, Week 7, Week 10) starting on Day 1, plus 960 mg vemurafenib orally twice daily throughout combination treatment.
- 720 mg Vemurafenib: These participants were receiving 720 mg vemurafenib in the Lead in Period prior to starting ipilimumab but after the dose limiting toxicities (DLTs) were identified, ipilimumab was not started. Due to disease stabilization, they continued on 720 mg vemurafenib alone orally twice daily.
- Total: Total of all reporting groups
Arm/Group | 3 mg/kg Ipilimumab + 960 mg Vemurafenib | 3 mg/kg Ipilimumab + 720 mg Vemurafenib | 720 mg Vemurafenib | Total
Number analyzed (Participants) | 6 | 4 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 1 | 8
  >=65 years | 3 | 0 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 6
  Male | 3 | 2 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 5 | 4 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: During the Lead In Period: Number of Participants With Adverse Events (AEs), AEs Leading to Drug Discontinuation, Serious Adverse Events (SAEs), and Deaths in Participants Treated With Vemurafenib Alone
Description: AEs graded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling, Gr 5=Death. Related=relationship to study drug reported as certain, probable, possible, or missing. Immune-related AEs (irAEs) characterized by potential association with inflammation and considered by investigator as drug related. Lead In Period: between the first vemurafenib dose and the day prior to the first ipilimumab dose.
Time Frame: From first vemurafenib dose to day prior to first ipilimumab dose (28 days); Patients who never progressed from Lead-in to combination treatment (720 mg Alone): first dose to last dose + 90 days (approximately 2 years)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- 960 mg Vemurafenib Lead in Period: Lead In Period: 28 Days of 960 mg vemurafenib orally twice daily (starting Day -27 or -13).
  Events between the first vemurafenib dose and the day prior to the first ipilimumab dose.
- 720 mg Vemurafenib Lead in Period: Lead In Period: 28 Days of 720 mg vemurafenib orally twice daily (starting Day -27 or -13).
  Events between the first vemurafenib dose and the day prior to the first ipilimumab dose.
- 720 mg Vemurafenib Alone: These participants were receiving 720 mg vemurafenib in the Lead in Period prior to starting ipilimumab but after the DLTs were identified, ipilimumab was not started. Due to disease stabilization, they continued on 720 mg vemurafenib alone orally twice daily.
  Events from first day of vemurafenib to last day of treatment + 90 days, up to date of data cut off for Primary Endpoint.
Arm/Group | 960 mg Vemurafenib Lead in Period | 720 mg Vemurafenib Lead in Period | 720 mg Vemurafenib Alone
Number analyzed (Participants) | 6 | 4 | 2
participants
  Deaths | 0 | 0 | 0
  Deaths due to disease progression | 0 | 0 | 0
  Grade 3 SAEs | 2 | 1 | 1
  Grade 4 SAEs | 0 | 0 | 0
  Grade 5 SAEs | 0 | 0 | 0
  Drug Related Grade 3 SAEs | 2 | 1 | 1
  Drug Related Grade 4 SAEs | 0 | 0 | 0
  AEs Leading to Study Drug Discontinuation | 0 | 0 | 0
  Grade 1 irAEs | 2 | 3 | 0
  Grade 2 irAEs | 1 | 0 | 0
  Grade 3 irAEs | 2 | 0 | 1
  Grade 4 irAEs | 0 | 0 | 0
  Grade 1 AEs | 0 | 1 | 0
  Grade 2 AEs | 2 | 2 | 0
  Grade 3 AEs | 4 | 1 | 2
  Grade 4 AEs | 0 | 0 | 0
  Grade 5 AEs | 0 | 0 | 0
  Drug Related Grade 1 AEs | 1 | 1 | 0
  Drug Related Grade 2 AEs | 2 | 2 | 0
  Drug Related Grade 3 AEs | 3 | 1 | 2
  Drug Related Grade 4 AEs | 0 | 0 | 0

2. Primary Outcome: During the Combination Treatment Period: Number of Participants With Adverse Events (AEs), AEs Leading to Drug Discontinuation, Serious Adverse Events (SAEs), and Deaths in Participants Treated With Concurrent Ipilimumab and Vemurafenib
Description: AEs graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling, Gr 5=Death. Related=relationship to study drug reported as certain, probable, possible, or missing. AEs: onset on or after ipilimumab start and within 90 days of last dose. Immune-related AEs (irAEs) characterized by potential association with inflammation and considered by investigator as drug related. Day 1=first dose of ipilimumab.
Time Frame: Combination drugs: Day 1 to last dose of drug + 90 days (approximately 2 years)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- 3 mg/kg Ipilimumab + 960 mg Vemurafenib: 3 mg/kg ipilimumab intravenously once every 3 weeks for 4 weeks (Week 1, Week 4, Week 7, Week 10) starting on Day 1 plus 960 mg vemurafenib orally twice daily and continuing during combination treatment.
- 3 mg/kg Ipilimumab + 720 mg Vemurafenib: 3 mg/kg ipilimumab intravenously once every 3 weeks for 4 weeks (Week 1, Week 4, Week 7, Week 10) starting on Day 1 plus 720 mg vemurafenib orally twice daily continuing during combination treatment.
Arm/Group | 3 mg/kg Ipilimumab + 960 mg Vemurafenib | 3 mg/kg Ipilimumab + 720 mg Vemurafenib
Number analyzed (Participants) | 6 | 4
participants
  Deaths | 4 | 1
  Deaths due to disease progression | 4 | 1
  Grade 3 SAEs | 3 | 2
  Grade 4 SAEs | 0 | 0
  Grade 5 SAEs | 2 | 0
  Drug Related Grade 3 SAEs | 5 | 2
  Drug Related Grade 4 SAEs | 0 | 0
  AEs Leading to Study Drug Discontinuation | 2 | 1
  Grade 1 irAEs | 1 | 0
  Grade 2 irAEs | 1 | 2
  Grade 3 irAEs | 4 | 2
  Grade 4 irAEs | 0 | 0
  Grade 1 AEs | 0 | 0
  Grade 2 AEs | 1 | 2
  Grade 3 AEs | 3 | 2
  Grade 4 AEs | 0 | 0
  Grade 5 AEs | 2 | 0
  Drug Related Grade 1 AEs | 0 | 0
  Drug Related Grade 2 AEs | 1 | 2
  Drug Related Grade 3 AEs | 5 | 2
  Drug Related Grade 4 AEs | 0 | 0

3. Primary Outcome: Number of Participants With Hepatic Dose Limiting Toxicities (DLT) in Participants Treated With Concurrent Ipilimumab and Vemurafenib
Description: DLT defined as a >= Grade 3 drug-related AE during induction with ipilimumab in combination with vemurafenib excluding: Grade 3 AE of tumor flare (defined as local pain, irritation, or rash localized at sites of known or suspected tumor); Grade 3 cutaneous squamous cell carcinoma; Grade 3 photosensitivity that resolved to a Grade 1 or baseline within 15 days; Grade 3 immune-mediated events of the skin (rash, pruritis) or endocrine systems (hypothyroidism, hyperthyroidism, hypopituitarism, adrenal insufficiency, hypogonadism and cushingoid) that resolved to a Grade 1 or baseline within 28 days; a transient (resolving within 6 hours of onset) Grade 3 infusion-related AE. Hepatic=elevated aspartate aminotransferase and alanine aminotransferase. Maximum tolerable dose (MTD) was defined as the maximum dose of combination treatment that could be given to 6 subjects such that no more than 2 subjects experience DLT. Day 1=first day of concurrent therapy with ipilimumab and vemurafenib.
Time Frame: Day 1 to last dose of drug + 90 (approximately 2 years)
Population: All participants who received at least one dose of concurrent study drugs.
Measure: Number; unit: participants
Groups:
- 3 mg/kg Ipilimumab + 960 mg Vemurafenib: 3 mg/kg ipilimumab intravenously once every 3 weeks for 4 weeks (Week 1, Week 4, Week 7, Week 10) starting on Day 1 plus 960 mg vemurafenib orally twice daily continuing during combination treatment.
Arm/Group | 3 mg/kg Ipilimumab + 960 mg Vemurafenib | 3 mg/kg Ipilimumab + 720 mg Vemurafenib
Number analyzed (Participants) | 4 | 2
participants | 4 | 2

ADVERSE EVENTS:
Time Frame: From the first vemurafenib dose in the Lead In Period to the last dose of combination drugs in the Treatment Period + 90 days, up to last patient, last visit, approximately 2 years.
Description: Final safety follow-up was 23 December 2013.
Groups:
- Lead-In Period 960 mg Vemurafenib: Lead In Period: 28 Days of 960 mg vemurafenib orally twice daily (starting Day -27 or -13).
  Events between the first vemurafenib dose and the day prior to the first ipilimumab dose.
- Lead-In Period 720 mg Vemurafenib: Lead In Period: 28 Days of 720 mg vemurafenib orally twice daily (starting Day -27 or -13).
  Events between the first vemurafenib dose and the day prior to the first ipilimumab dose.
- Lead- In Period 720 mg Vemurafenib Alone: These participants were receiving 720 mg vemurafenib in the Lead in Period prior to starting ipilimumab but after the DLTs were identified, ipilimumab was not started. Due to disease stabilization, they continued on 720 mg vemurafenib alone orally twice daily.
Arm/Group | Lead-In Period 960 mg Vemurafenib | Lead-In Period 720 mg Vemurafenib | Lead- In Period 720 mg Vemurafenib Alone | 3 mg/kg Ipilimumab + 960 mg Vemurafenib | 3 mg/kg Ipilimumab + 720 mg Vemurafenib
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/4 | 1/2 | 5/6 | 2/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 2/2 | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-In Period 960 mg Vemurafenib (N=6) | Lead-In Period 720 mg Vemurafenib (N=4) | Lead- In Period 720 mg Vemurafenib Alone (N=2) | 3 mg/kg Ipilimumab + 960 mg Vemurafenib (N=6) | 3 mg/kg Ipilimumab + 720 mg Vemurafenib (N=4)
Cytomegalovirus enteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 4 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-In Period 960 mg Vemurafenib (N=6) | Lead-In Period 720 mg Vemurafenib (N=4) | Lead- In Period 720 mg Vemurafenib Alone (N=2) | 3 mg/kg Ipilimumab + 960 mg Vemurafenib (N=6) | 3 mg/kg Ipilimumab + 720 mg Vemurafenib (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 3
Oedema peripheral (General disorders) | 0 | 0 | 0 | 3 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 2
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Episcleritis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 3 | 0 | 1 | 0 | 3
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 4 | 3
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 2
Coordination abnormal (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 1
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 3 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 2
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
In Phase 1 of the study, MTD was not reached because more than 2 of 6 treated participants experienced DLTs with the combination therapy. Enrollments in Phase 1 were terminated and Phase 2 was not started so only overall safety was summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.